CLINICAL TRIAL: NCT03300882
Title: Prospective Multicenter Cytomegalovirus (CMV) Specific Immune Monitoring to Predict Patient Risk After Lung Transplantation (CTOT-22)
Brief Title: PREDICT Cytomegalovirus (CMV)
Acronym: PREDICT CMV
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOT-22; NIAID CRMS ID#: 38277 (Other: DAIT NIAID)
Record Dates: First submitted 2017-09-25; First posted 2017-10-04 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Lung Transplant
Keywords: Study co-enrollment (CTOT-20 and CTOT-22); cytomegalovirus (CMV); CMV seropositive positive recipient; CMV infection; CMV-specific immunity; immunologic monitoring
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Methods; Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells (PBMCs) and plasma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CMV+ First Lung Transplant Recipients: Participants enrolled in one of four North American sites in clinical research study CTOT-20 (Clinical Trials.gov ID: NCT02631720) who are cytomegalovirus positive by serology (e.g., CMV Recipient positive).
  Interventions: Other: Procedure

INTERVENTIONS:
Other: Procedure — Serial blood draws. Participants will be enrolled either pre-transplant or within 45 days post-transplant and will be followed over the course of 18 months post transplant. Protocol mandated serial measurement of cytomegalovirus (CMV)-specific immune signature will occur pre-transplant (as applicable) and at post-transplant timepoint months 2, -3, -6, -9, -12 and -18.
  Other Names: Serial blood draws; Phlebotomy; Venipuncture

SUMMARY:
The overall objective of this study is to establish a personalized test to measure individualized cytomegalovirus (CMV) specific immunity in lung transplant recipients in an effort to guide antiviral prophylaxis duration in clinical practice.

Targeted participants are those:

* enrolled in clinical research study CTOT-20 (Clinical Trials.gov ID: NCT02631720) who
* are CMV recipient positive by serology as determined using methods in accordance with current local organ procurement organization policies.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is a common virus. The virus is spread from one person to another through infected body fluids. In those with a normal immune system, CMV does not cause much of a problem. The immune system keeps the virus under control so most people do not have any symptoms. Once infected, the virus usually stays dormant (inactive) in the body for a person's entire life. This means some of the cells in the body are infected and the virus can become active again.

Lung transplant recipients take anti-rejection medicines to prevent the body from rejecting the transplanted lung(s). Although anti-rejection medications help protect the transplanted lung(s) from the body's immune system, these medications also decrease the body's ability to fight infections. This reduces the immune system's ability to control viruses like CMV. Many transplant recipients take an antiviral medication early after transplant to help the body control the CMV virus. This is the time that risk of infection would be highest. Sometimes recipients get an active CMV infection after stopping these medicines. If this happens, the infection is treated and monitored.

In this study, investigators are trying to determine whether a blood test can predict development of active CMV infection in lung transplant recipients. Specifically, the clinical research study will prospectively assess the performance of an immune signature based on the "ex vivo" measurement of T cell CMV specific immunity in predicting freedom from future CMV infections among recipient positive (R+) lung transplant participants receiving standard durations of valganciclovir prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

* Must be able to understand and provide written informed consent;
* Anticipated listing for lung transplantation OR listed for lung transplant OR is within 45 days of having received a single or bilateral cadaveric donor lung transplant;
* Undergoing first lung transplant operation;
* Transplant surgery to be performed or performed at enrolling center;
* Concurrent participation in CTOT-20 (Clinical Trials.gov ID: NCT02631720); and
* CMV-seropositive lung transplant recipient, using methods in accordance with current local organ procurement organization policies.

  * Note: Concurrent participation in immune monitoring studies or interventional device trials are permitted.

Exclusion Criteria:

Individuals who meet any of the following criteria are not eligible for enrollment as study participants:

* Unwilling to enroll in CTOT-20 (Clinical Trials.gov ID: NCT02631720);
* Multi-organ recipient;
* Prior recipient of any solid organ transplant, including prior lung transplant;
* Prior or concurrent recipient of bone marrow transplant;
* Human Immunodeficiency Virus (HIV) infection;
* Pregnant or planned pregnancy;
* Any condition that, in the investigator's opinion, would make it unlikely for the recipient to complete follow up procedures or complete the study; or
* Participation in an investigational drug trial at the time of enrollment visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult lung transplant recipients undergoing lung transplant at one of the four participating centers and concurrently enrolled in CTOT-20 (Clinical Trials.gov ID: NCT02631720).
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Time from CMV Prophylaxis Discontinuation Post-Transplant to First Detection of CMV Infection or CMV Disease within 6 months Post CMV Prophylaxis Discontinuation | From CMV Prophylaxis Discontinuation to 6 Months Post CMV Prophylaxis Discontinuation
  Participants will be evaluated for CMV infection or disease according to each center's standard of care clinical protocol. All centers have aligned their clinical practice to include, at a minimum, a CMV infection and a CMV disease assessment at the time of prophylaxis discontinuation, monthly for the first 6 months after discontinuation, and quarterly after that up to 18 months post transplantation.
Time from CMV Prophylaxis Discontinuation Post-Transplant to First Detection of CMV Infection or CMV Disease Within 18 Months Post-Transplant | From CMV Prophylaxis Discontinuation to 18-Months Post-Transplant
  Participants will be evaluated for CMV infection or disease according to each center's standard of care clinical protocol. All centers have aligned their clinical practice to include, at a minimum, a CMV infection and a CMV disease assessment at the time of prophylaxis discontinuation, monthly for the first 6 months after discontinuation, and quarterly after that up to 18 months post transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Snyder, MD, MHS, Study Chair — Duke University Medical Center: Transplantation; Scott Palmer, MD, MHS, Study Chair — Duke University Medical Center: Transplantation
Locations (4):
- United States (3):
  - Johns Hopkins Hospital: Transplantation, Baltimore, Maryland
  - Duke University Medical Center: Transplantation, Durham, North Carolina
  - Cleveland Clinic Foundation: Transplantation, Cleveland, Ohio
- Toronto General Hospital: Transplantation, Toronto, Canada

REFERENCES:
- [Background] Snyder LD, Chan C, Kwon D, Yi JS, Martissa JA, Copeland CA, Osborne RJ, Sparks SD, Palmer SM, Weinhold KJ. Polyfunctional T-Cell Signatures to Predict Protection from Cytomegalovirus after Lung Transplantation. Am J Respir Crit Care Med. 2016 Jan 1;193(1):78-85. doi: 10.1164/rccm.201504-0733OC. PMID 26372850
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Clinical Trials in Organ Transplantation (CTOT) — http://www.ctotstudies.org/